CLINICAL TRIAL: NCT00001929
Title: NMDA-Receptor Blockade With Eliprodil in Parkinson's Disease
Brief Title: Treatment of Parkinson's Disease With Eliprodil
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 990078; 99-N-0078
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-01

CONDITIONS: Movement Disorders; Parkinson Disease
Keywords: Dyskinesias; Glutamate Antagonist; Levodopa
MeSH Terms: conditions — Movement Disorders; Parkinson Disease; Dyskinesias | interventions — eliprodil

INTERVENTIONS:
Drug: Eliprodil

SUMMARY:
Patients with Parkinson's disease are missing the chemical neurotransmitter dopamine. This occurs as a result of destructive changes in an area of the brain responsible for making dopamine, the basal ganglia. Patients with the disease experience, rigid muscles, stooped posture, and a shuffling-type walk (gait).

In this study researchers plan to evaluate the effectiveness of the drug eliprodil for the treatment of Parkinson's Disease. Eliprodil works by blocking special receptors (NMDA) that are associated with the symptoms of Parkinson's Disease.

DETAILED DESCRIPTION:
The objectives of this study are to evaluate the acute effects of the NR2B subtype-selective NMDA antagonist eliprodil on levodopa-associated motor response complications in patients with advanced Parkinson's Disease (PD).

ELIGIBILITY:
All patients will carry a diagnosis of idiopathic Parkinson's Disease based on the presence of a characteristic clinical history and neurologic findings. Most will have relatively advanced disease with associated motor response complications.

Males and females between the ages of 18-75.

No presence or history of any medical condition that can reasonably be expected to subject the patient to unwarranted risk.

No patients with baseline QTc prolongation (greater than 440 msec).

No pregnant women nor those not practicing effective means of birth control.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 1999-03; Study Completion 2001-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bergman H, Wichmann T, DeLong MR. Reversal of experimental parkinsonism by lesions of the subthalamic nucleus. Science. 1990 Sep 21;249(4975):1436-8. doi: 10.1126/science.2402638.
- [Background] Mitchell IJ, Clarke CE, Boyce S, Robertson RG, Peggs D, Sambrook MA, Crossman AR. Neural mechanisms underlying parkinsonian symptoms based upon regional uptake of 2-deoxyglucose in monkeys exposed to 1-methyl-4-phenyl-1,2,3,6-tetrahydropyridine. Neuroscience. 1989;32(1):213-26. doi: 10.1016/0306-4522(89)90120-6. PMID 2586750